CLINICAL TRIAL: NCT03443609
Title: Diagnostic Multicenter Phase II Study, Prospective, Comparative, of 68Ga-HBED-PSMA PET / CT and Conventional Imaging Procedures in Occult Biological Relapse Prostate Cancer
Brief Title: Study of 68Ga-HBED-PSMA PET/CT and Conventional Imaging in Occult Biological Relapse Prostate Cancer
Acronym: PSMA REBIOLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-N-2016-01
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer Recurrent
Keywords: occult prostate cancer recurrence; PSA; 68Ga-HBED-CC-PSMA PET / CT

STUDY DESIGN:
Intervention Model Description: All the imaging sequences will be done in an outpatient setting. There will be no premedication or other treatment before and after 68Ga-HBED-CC-PSMA PET scans. PET / CT will be performed at participating centers on a hybrid PET camera.
  68Ga-HBED-CC-PSMA will be administered to the patient by single intravenous injection (Y-infused with isotonic saline infusion) within 60 min of reconstitution of the radiopharmaceutical.
  The first TEP 68Ga-HBED-CC-PSMA whole body acquisition starts 60 min after the injection of 150 MBq of 68Ga-HBED-CC-PSMA and continues for 20-30 minutes, the second full-body acquisition of the same duration takes place 120 minutes after the injection is a total duration of 1 hour of imaging and 2:30 to 3:00 in the service.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-HBED-CC-PSMA PET / CT (Other): Patients will receive 68Ga-HBED-CC-PSMA PET / CT imaging for the detection of prostate cancer recurrence sites. This determination will be made at the "patient" and "lesion" level by reference to the gold standard (or truth standard) that will be obtained from the histology data and / or from an imaging and evolution follow-up. PSA over a period of at least 6 months (RECIST 1.1 criteria).
  Interventions: Diagnostic Test: 68Ga-HBED-CC-PSMA PET / CT

INTERVENTIONS:
Diagnostic Test: 68Ga-HBED-CC-PSMA PET / CT — Patient will receive a specific PET / CT with PSMA

SUMMARY:
68Ga-HBED-CC-PSMA is a radiopharmaceutical allowing a new imaging modality for the detection of prostate cancer recurrences, used in recent years in clinical studies by some teams mainly in Europe (1-6 ).

The aim of this study is to study the diagnostic performance of 68Ga-HBED-PSMA PET / CT in occult recurrent carcinoma (PCa) by prospectively comparing it to the standard techniques used in this indication: optimized bone scintigraphy with double TEMP / CT systematic and abdominopelvic MRI. The therapeutic impact and tolerance of this examination will also be evaluated.

The expected results are a demonstration of the superiority of 68Ga-HBED-PSMA PET compared to the standard assessment, with a potential impact on the therapeutic management of patients

DETAILED DESCRIPTION:
METHODOLOGY:

Phase II imaging study, prospective, multicenter non-randomized.

MAIN OBJECTIVE:

To determine the added value of 68Ga-HBED-CC-PSMA PET / CT in imaging investigations in terms of the sensitivity of detection of biologic suspected prostate cancer recurrence site locations on the elevation of plasma PSA, while all conventional imaging exams are negative or questionable ("occult recurrence")

SECONDARY OBJECTIVE:

* Evaluate the clinical impact of 68Ga-HBED-CC-PSMA PET / CT in imaging exam by the predicted rate of change in therapeutic attitude.
* Evaluate the relevance of decisions made after PET / CT 68Ga-HBED-CC-PSMA.
* Determine the added value of 68Ga-HBED-CC-PSMA PET / CT in terms of specificity and predictive value for detecting secondary locations. This determination will be at the "patient" level and at the "lesion" level
* To determine the added value of the 2nd PET / CT at 68Ga-HBED-CC-PSMA (2h after the radiopharmaceutical injection) in terms of specificity and predictive value for the detection of secondary locations in relation to the added value of the 1st PET / CT acquisition at 68Ga-HBED-CC-PSMA. This determination will be at the "patient" level and at the "lesion" level.
* Confirm the perfect tolerance of 68Ga-HBED-CC-PSMA.

STUDY PROCEDURE :

All the imaging sequences will be done in an outpatient setting. There will be no premedication or other treatment before and after 68Ga-HBED-CC-PSMA PET scans. PET / CT will be performed at participating centers on a hybrid PET camera.

68Ga-HBED-CC-PSMA will be administered to the patient by single intravenous injection (Y-infused with isotonic saline infusion) within 60 min of reconstitution of the radiopharmaceutical.

The first TEP 68Ga-HBED-CC-PSMA whole body acquisition starts 60 min after the injection of 150 MBq of 68Ga-HBED-CC-PSMA and continues for 20-30 minutes, the second full-body acquisition of the same duration takes place 120 minutes after the injection is a total duration of 1 hour of imaging and 2:30 to 3:00 in the service.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Diagnosis of histologically proven prostate cancer.
3. Patient having benefited from previous curative treatment (prostatectomy, radiotherapy, ultrasound, cryotherapy ...), with a significant decrease in the plasma concentration of PSA at the end of treatment (= indisputable PSA)
4. Biologic recurrence documented by abnormal results in 2 assays of plasma PSA concentration in the same laboratory.
5. Value of the plasma concentration of the last PSA assay during the 4 months preceding D0: 0.05 ng / mL ≤ PSA <1.6 ng / mL
6. Conventional imaging assessment already carried out, including at least one optimized skeleton scintigraphy with thoracoabdominopelvic TEMP / CT (or 18F-Choline TEP) and pelvic MRI (or abdominopelvic CT if contraindicated MRI) less than 6 weeks old. All of these tests must have been interpreted as "negative" or "questionable" (without "suggestive" or "suspect" aspects of malignancy) written by the imaging specialist.
7. Karnofsky ≥ 70 or ECOG 0-1
8. Life expectancy of at least 6 months
9. The patient has given his written consent.
10. Patient affiliated to a social security scheme

Exclusion Criteria:

1. Another progressive cancerous condition, except for basal cell cancers.
2. Acute inflammatory condition,
3. Implementation of treatment (eg chemotherapy) or change of treatment (eg hormone therapy) since skeletal scintigraphy, abdominopelvic MRI or the last serum PSA test.
4. Radiotherapy, chemotherapy or other anti-tumor treatment during the 6 weeks preceding PET,
5. Agitation; impossibility to hold motionless for at least 1 hour, or known claustrophobia
6. Poor predictable compliance or inability to undergo medical follow-up of the test for geographical, social or psychological reasons,
7. Intellectual inability to sign informed consent
8. Persons deprived of liberty or guardianship (including trusteeship),

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
added value of 68Ga-HBED-CC-PSMA PET / CT in imaging examinations in terms of detection sensitivity of recurrence sites | 6 months
  To determine the added value of 68Ga-HBED-CC-PSMA PET / CT in imaging examinations in terms of detection sensitivity of prostate cancer recurrence sites, biologically suspected of elevated plasma concentrations of PSA, while all conventional imaging tests are negative or questionable: "occult recurrence".

CONTACTS AND LOCATIONS:
Overall Officials: ROUSSEAU Caroline, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- ICO René Gauducheau, Saint-Herblain, France

REFERENCES:
- [Derived] Rousseau C, Le Thiec M, Ferrer L, Rusu D, Rauscher A, Maucherat B, Frindel M, Baumgartner P, Fleury V, Denis A, Morel A, Varmenot N, Debeaupuis E, Campion L, Kraeber-Bodere F. Preliminary results of a 68 Ga-PSMA PET/CT prospective study in prostate cancer patients with occult recurrence: Diagnostic performance and impact on therapeutic decision-making. Prostate. 2019 Sep;79(13):1514-1522. doi: 10.1002/pros.23869. Epub 2019 Aug 17. PMID 31421657